CLINICAL TRIAL: NCT06368310
Title: First in Human (FIH) Clinical Investigation of Safety and Feasibility of a Novel Graphene Micro-electrocorticography Array for Brain Mapping in Neuro-oncology
Brief Title: FIH Clinical Investigation of Graphene Electrodes for Brain Mapping
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Northern Care Alliance NHS Foundation Trust (Other); European Commission (Other); Inbrain Neuroelectronics (Industry)
Responsible Party: Principal Investigator, David Coope, Academic Consultant in Neurosurgery, Northern Care Alliance NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: R124807; 23/WM/0166 (Other: NHS Research Ethics Committee Reference)
Record Dates: First submitted 2024-03-20; First posted 2024-04-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Brain Tumor; Glioma
Keywords: Electrocorticography; Subdural electrode; Graphene
MeSH Terms: conditions — Brain Neoplasms; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Patients with suspected gliomas (intrinsic primary brain tumors) in whom surgical resection under general anesthesia with neurophysiological monitoring or under awake conditions where language mapping is planned.
  Interventions: Device: INBRAIN Graphene Cortical Interface

INTERVENTIONS:
Device: INBRAIN Graphene Cortical Interface — Study device to be evaluated intra-operatively alongside standard of care neurophysiological monitoring.

SUMMARY:
The goal of this clinical investigation of a medical device is to test the safety of graphene based electrodes when used during surgery for resection of brain tumors. The main questions that it aims to answer are:

* To understand the safety of the Graphene Cortical Interface when used during brain tumor surgery (primary objective);
* To assess the quality of the brain signals recorded with the Graphene Cortical Interface, their ability to stimulate the brain, how stable their function is over the duration of an operation, and their suitability for use in the operating theatre (secondary objectives).

Participants will undergo tumor surgery as usual with the study electrodes being tested alongside a standard monitoring system. If they are awake for part of their surgery they may be asked to complete specific tasks such as naming objects from a list modified for the study, to evaluate the capability to decode brain signals (exploratory objective). They will be monitored subsequently for any complications including undergoing an additional MRI scan 6 weeks after their surgery.

DETAILED DESCRIPTION:
During surgical operations within the brain such as the removal of a tumor, electrodes are commonly used to map specific brain functions or monitor brain activity. These are most commonly flexible plastic devices with embedded metallic contacts that allow electrical activity in the brain to be detected and measured. They may also be used to stimulate precise areas of the brain to either trigger or block a response such as the contraction of a muscle. This allows the surgeon to define which regions of the brain are involved in controlling critical functions such as movement or speech so that these areas can be protected during the operation.

There remain limitations with the design and physical characteristics of commercially available electrodes for use during brain operations. These include the limited ability of conventional materials to fold over the complex shape of the brain and the need to use comparatively large metallic contacts to detect the tiny electrical signals. This study will be the first to introduce a new generation of electrodes which have been designed to overcome these limitations. They are extremely thin and flexible allowing them to follow the surface of the brain and to be used in locations within and around the brain for which the standard electrodes are unsuitable. The contact surfaces that detect electrical activity and enable and stimulate the brain have been replaced with graphene which is a novel carbon-based material. The use of graphene allows electrodes to be made that are more sensitive to the tiny electrical signals of the brain. This means that they can be much smaller and closer together providing increased detail in the recording and potentially enabling signals to be detected that would previously have required such long recordings that they could not be used to guide decision making during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Solitary supratentorial tumor radiologically consistent with glioma (intrinsic primary brain tumor) on standard diagnostic MRI;
* Planned for surgery under awake conditions or under general anesthesia with intra-operative electrocorticography (ECoG);
* English as first language for those subjects with tumors associated with language areas;
* Karnofsky performance score > 70 and World Health Organization (WHO) performance status score ≤ 1;
* Willing and able to understand and provide informed consent for participating in the study.

Exclusion Criteria:

* Contraindications to magnetic resonance imaging (e.g., incompatible implanted devices);
* Previous cranial surgery or radiotherapy;
* Subjects expected to undergo craniotomy of less than 5 cm in maximum diameter (bone to bone)
* Known extracranial malignant neoplasm;
* Pregnant or lactating women;
* Renal impairment sufficient to limit Gadolinium administration (EGFR <60 ml/min)
* For those subjects with tumors associated with language areas, any contraindication which could preclude them from performing the whole awake intra operative tasks at the discretion of the Investigator (e.g., language function not suitable for monitoring tasks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-03-21 (Estimated); Study Completion 2026-03-21 (Estimated)

PRIMARY OUTCOMES:
To evaluate the preliminary safety of the investigational device for its intended use | Through study completion, an average of 3 months
  All adverse events (including, but not limited to, adverse device events)

SECONDARY OUTCOMES:
Assess the ability of the device to record signals from the brain | During surgical procedure
  Performance of detecting signals from the brain by sensing of electrical brain activity
Evaluate the ability of the device to provide functional stimulation of the brain | During surgical procedure
  Performance of functional stimulation of the brain by inducing evoked motor responses measured as peripheral muscle electromyography (EMG)
Assess stability of sensing and stimulating electrodes | During surgical procedure
  Stability of electrodes by evaluation of impedance measurements over time
Evaluate device usability - an assessment by questionnaire of the operating surgeon's impression of the suitability of the device for sensing and stimulation during brain tumor surgery | During surgical procedure
  Study specific questionnaire to be completed by the operating surgeon including ease of handling, positioning and removal of the electrode. The study specific 'Device Usability' tool scores outcomes on a scale of 1-4 where 4 represents a favourable feature.

OTHER OUTCOMES:
Assess the quality of the recorded somatosensory evoked potentials (SEPs) - sensing part A (exploratory) | During surgical procedure
  Assessing the quality of recorded brain activity by measuring signal to noise ratio (SNR) during stimulation of a peripheral nerve
Assess the quality of the recorded baseline brain activity - sensing part B (exploratory) | During surgical procedure
  Assessing the quality of recorded brain activity at rest (or under anaesthesia) evaluated as the power spectral density (PSD)
Assess the ability of detecting brain evoked responses during stimulation of the brain (exploratory) | During surgical procedure
  Preliminary assessment of the ability of the device to detect changes in brain activity evoked in response to stimulation of distant but connected brain regions
Evaluate decoding capability from data recorded during language task (exploratory) | During surgical procedure
  Preliminary evaluation of the ability to detect changes in brain activity that correspond to word or sound generation as the participant completes a standardized object naming task (quantified by classification accuracy)
Evaluate signal characteristics of tumour infiltrated brain regions (exploratory) | During surgical procedure
  Preliminary evaluation of changes in the pattern of brain activity in healthy brain versus that infiltrated by tumour quantified by changes in the power spectral density (PSD)

CONTACTS AND LOCATIONS:
Overall Officials: David J Coope, PhD FRCS, Principal Investigator — Northern Care Alliance NHS Foundation Trust
Locations (1):
- Manchester Centre for Clinical Neurosciences, Northern Care Alliance NHS Foundation Trust, Salford, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Viana D, Walston ST, Masvidal-Codina E, Illa X, Rodriguez-Meana B, Del Valle J, Hayward A, Dodd A, Loret T, Prats-Alfonso E, de la Oliva N, Palma M, Del Corro E, Del Pilar Bernicola M, Rodriguez-Lucas E, Gener T, de la Cruz JM, Torres-Miranda M, Duvan FT, Ria N, Sperling J, Marti-Sanchez S, Spadaro MC, Hebert C, Savage S, Arbiol J, Guimera-Brunet A, Puig MV, Yvert B, Navarro X, Kostarelos K, Garrido JA. Nanoporous graphene-based thin-film microelectrodes for in vivo high-resolution neural recording and stimulation. Nat Nanotechnol. 2024 Apr;19(4):514-523. doi: 10.1038/s41565-023-01570-5. Epub 2024 Jan 11. PMID 38212522
- See also: European Union Graphene Flagship — https://graphene-flagship.eu/about/first-10-years/core-3-work-packages/work-package-5-biomedical-technologies/